CLINICAL TRIAL: NCT05043714
Title: A Multicentre, Open-label, Non-randomized, Phase 1a/1b Study of NG-641, a Tumour-selective and Transgene-expressing Adenoviral Vector, in Combination With Nivolumab (or Standard of Care PD-1 Inhibition) in Patients With Metastatic or Advanced Epithelial Tumours (NEBULA)
Brief Title: Study of NG-641 in Combination With Nivolumab in Metastatic or Advanced Epithelial Tumours
Acronym: NEBULA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NG-641-03
Record Dates: First submitted 2021-09-02; First posted 2021-09-14 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Cancer; Epithelial Tumor
Keywords: Metastatic Cancer; Epithelial Tumor; Viral vector; Advanced; PsiOxus
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous (Experimental): Phase 1a Part A: One cycle (28 days) of NG-641 on Days 1, 3 and 5 and nivolumab on Day 15, followed by nivolumab every 4 weeks.
  Phase 1a Part B: NG-641 on Days 1, 3 and 5 and one nivolumab on Day 15 in each of up to eight 28-day cycles.
  Interventions: Biological: NG-641 in combination with Nivolumab

INTERVENTIONS:
Biological: NG-641 in combination with Nivolumab — NG-641 is a replication competent adenoviral vector producing a bispecific T cell activator (TAc) targeting fibroblast activation protein (FAP) plus immune enhancer genes CXCL9/CXCL10/IFNa2. This can lead to killing of tumor cells and stimulation of immunity against the tumor cells.
  Nivolumab is a human monoclonal antibody that targets the PD-1 cluster of differentiation 279 cell surface membrane receptor.

SUMMARY:
This is a phase 1a/1b, multicentre, open-label, non-randomized study of NG-641 in combination with nivolumab (or standard of care PD-1 inhibition) in patients with metastatic or advanced epithelial tumours.

The purpose is to characterize the safety and tolerability of NG-641 in combination with nivolumab in patients with metastatic or advanced epithelial tumours and to determine the recommended dose of NG-641 in combination with nivolumab for further development in patients with metastatic or advanced epithelial tumours

DETAILED DESCRIPTION:
The Phase 1a part of the study is a dose escalation phase and is composed of two parts: Part A, which is investigating NG-641 administration (single cycle) by intravenous (IV) infusion in combination with up to 8 cycles of nivolumab; and Part B, which is investigating multicycle NG-641 administration (up to 8 cycles) by IV infusion in combination with up to 8 cycles of nivolumab. Both parts will include patients with metastatic or advanced tumours. Part B will open once a recommended starting dose of NG-641 is identified from the single-cycle dose escalation. Dose escalation in Part A may continue in parallel once Part B has opened.

The Phase 1b part of the study will further investigate the efficacy and safety of the selected dose regimen in up to three of the tumour types evaluated in phase 1b (tumour-specific Dose Expansion Cohorts A, B and C). A Simon 2-stage design will be used, with sample size calculations and futility criteria specific to each individual expansion cohort. Patients enrolled in Cohort A will have recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) that is considered incurable by local therapies and has been recently treated with a first-line platinum-based chemotherapy regimen or platinum-based chemotherapy plus pembrolizumab.

Patients enrolled in Cohort A will be subdivided in to two groups according to whether they have received prior anti-PD-1 therapy (Cohort A1, chemotherapy regimen without pembrolizumab; Cohort A2, chemotherapy regimen with pembrolizumab) with each sub-cohort using a separate Simon 2-stage model. Patients in Cohort A2 who are already receiving pembrolizumab as standard of care at enrolment may continue this background treatment in combination with the recommended NG-641 dose; patients are permitted to switch to nivolumab at the Investigator's discretion. Cohorts B and C will be defined in a future protocol update that will be submitted for approval prior to these cohorts opening.

Following treatment, patients will be followed every 8 weeks until 12 months from first dose for disease status, overall survival, further cancer therapy and the best response and date of disease progression on further cancer therapy. These assessments may be performed by telephone calls or at routine visits to the hospital.

ELIGIBILITY:
Inclusion Criteria:

Phase 1a:

1. Patients must have histologically or cytologically documented metastatic/advanced epithelial cancer that has relapsed from or is refractory to standard treatment, or for which no standard treatment is available.
2. At least one measurable site of disease according to RECIST Version 1.1 criteria; this lesion must be either (i) outside a previously irradiated area or (ii) progressive if it is in a previously irradiated area
3. Tumour accessible for biopsy, biopsy deemed safe by the Investigator, and patient willing to consent to tumour biopsies

All patients:

1. Provide written informed consent to participate
2. Ability to comply with study procedures in the Investigator's opinion
3. Aged 18 years or over
4. ECOG performance status 0 or 1
5. Predicted life expectancy of ≥6 months
6. Adequate lung reserve
7. Adequate renal function
8. Adequate hepatic function
9. Adequate bone marrow function
10. Meeting reproductive status requirements

Exclusion Criteria

1. Prior or planned allogeneic or autologous bone marrow or organ transplantation
2. Splenectomy
3. Active infections requiring antibiotics, physician monitoring or systemic therapy within 1 week of the anticipated first dose of study drug, or recurrent fevers (>38.0˚C) associated with a clinical diagnosis of active infection
4. Treatment with the antiviral agents: ribavirin, adefovir, lamivudine, cidofovir or paxlovid within 10 days prior to the first dose of study treatment; or pegylated interferon in the 4 weeks before the first dose of study treatment
5. Known history of hepatitis B infection or known active hepatitis C infection . Known history of HIV infection
6. Patients who have active, known or suspected autoimmune disease that has required systemic therapy in the past 2 years, are immunocompromised in the opinion of the Investigator, or are receiving long-term systemic immunosuppressive treatment
7. Treatment with any live, live-attenuated or COVID-19 vaccine in the 30 days before the first dose of NG-641 or nivolumab
8. Treatment with any other vaccine (including known non-live/live-attenuated and non-adenoviral COVID-19 vaccines) in the 7 days before the first dose of NG-641
9. History of prior Grade 3-4 acute kidney injury or other clinically significant renal impairment
10. History of clinically significant interstitial lung disease or non-infectious pneumonitis
11. Lymphangitic carcinomatosis
12. Infectious or inflammatory bowel disease in the 3 months before the first dose of study treatment
13. Any known CTCAE Grade ≥2 coagulation abnormality/coagulopathy
14. Any clinically significant cardiovascular, peripheral vascular, cerebrovascular, or thromboembolic event in the 6 months before the first dose of study treatment
15. Grade 3 or 4 gastrointestinal bleeding (or risk factors for gastrointestinal bleeding), haemoptysis, or any history of bleeding requiring an investigative procedure, transfusion or hospitalisation in the 6 months before the first dose of study treatment
16. Tumour location/extent considered by the Investigator to present a significant risk if tumour flare or necrosis were to occur
17. Known retinopathy, including retinal haemorrhages, cotton wool spots, papilloedema, optic neuropathy and retinal artery or vein obstruction
18. Active clinically severe depression
19. Use of the following prior therapies/treatments

    * Treatment with any other enadenotucirev-based virus (parent virus or transgene-modified variants), or fibroblast activation protein (FAP) targeting agent at any time
    * Treatment with an investigational or licensed anti-cancer monoclonal antibody (mAb), immune checkpoint inhibitor, immune stimulatory treatment, or other biological therapy in the 28 days prior to the first dose of study treatment
    * Prior anti-PD-1/PD-L1 therapy is permitted without a 'washout' phase
    * Treatment with an investigational or licensed chemotherapy, targeted small molecule, or other investigational drug in the 14 days or five half-lives (whichever is shorter) before the first dose of study treatment
    * Major surgery in the 28 days before the first dose of study treatment
    * Radiation therapy in the 14 days before the first dose of study treatment
    * Treatment with complementary medications to treat the disease under study within the 14 days prior to first study treatment
    * Bisphosphonate therapy or treatment with Receptor Activator of Nuclear factor Kappa-Β (RANK)-ligand inhibitors for metastatic bone disease is permitted
20. All toxicities attributed to prior anti-cancer therapy (including radiation therapy) must have resolved to Grade 1 or baseline before the first dose of study treatment (see protocol for exceptions)
21. Known allergy or hypersensitivity (Grade ≥3) to NG-641 transgene, immune checkpoint inhibitor products or formulation, or other monoclonal antibodies
22. Known hypersensitivity to both cidofovir and valacyclovir
23. Discontinuation from prior treatment with an immune therapy due to a Grade ≥3 immune-related AE, or any history of life-threatening toxicity related to prior immune therapy except those that are unlikely to re-occur with standard countermeasures
24. Other prior malignancy active within the previous 3 year (see protocol for exceptions)
25. Symptomatic brain metastases or any leptomeningeal metastases that are symptomatic and/or requires treatment (see protocol for exceptions)
26. Any serious or uncontrolled medical disorder that, in the opinion of the Investigator or the Medical Monitor, may increase the risk associated with study participation or study treatment administration, impair the ability of the patient to receive protocol therapy or interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (safety and tolerability) in study of NG-641 in combination with nivolumab | 30 days after last dose of study drug
  Incidence of: adverse events (AEs), serious adverse events (SAEs), AEs leading to discontinuation of study treatment or study discontinuation and AEs resulting in death and Incidence of AEs meeting protocol defined dose-limiting toxicity (DLT) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ottensmeier, MD, Principal Investigator — Clatterbridge Cancer Centre
Locations (6):
- United States (4):
  - Providence Medical Foundation, Fullerton, California
  - UCLA Department of Medicine, Santa Monica, California
  - Moffitt-Advent Health Clinical Research Unit, Celebration, Florida
  - University of Cincinnati Cancer Center, Cincinnati, Ohio
- United Kingdom (2):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool, Lancashire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire

REFERENCES:
- [Derived] Khalil DN, Prieto Gonzalez-Albo I, Rosen L, Lillie T, Stacey A, Parfitt L, Soff GA. A tumor-selective adenoviral vector platform induces transient antiphospholipid antibodies, without increased risk of thrombosis, in phase 1 clinical studies. Invest New Drugs. 2023 Apr;41(2):317-323. doi: 10.1007/s10637-023-01345-8. Epub 2023 Mar 10. PMID 36897458